CLINICAL TRIAL: NCT00982826
Title: A Blinded, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profiles of Single and Multiple Doses (7 Days) of ABT-072 and an Open-label Study to Evaluate the Effect of Food on the Pharmacokinetic
Brief Title: Single and Multiple Dose Evaluation of ABT-072 and to Evaluate the Effect of Food on the Pharmacokinetics of ABT-072
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Barry Bernstein, Project Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: M11-057
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C
Keywords: Phase 1; Single and Multiple Ascending Dose; Food Effect
MeSH Terms: conditions — Hepatitis C | interventions — ABT-072

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): ABT-072 tablet single ascending dose
  Interventions: Drug: ABT-072
- 2 (Experimental): Placebo tablet
  Interventions: Drug: Placebo
- 3 (Experimental): ABT-072 tablet administered under non-fasting conditions.
  Interventions: Drug: ABT-072
- 4 (Experimental): ABT-072 tablet administered under fasting conditions
  Interventions: Drug: ABT-072
- 5 (Experimental): ABT-072 tablet multiple ascending dose
  Interventions: Drug: ABT-072

INTERVENTIONS:
Drug: ABT-072 — See Arms information for a detailed description.
  Arms: 1; 3; 4; 5
Drug: Placebo — See Arms information for a detailed description.
  Arms: 2

SUMMARY:
To assess the safety, tolerability and pharmacokinetics of the ABT-072 tablet formulation administered as a single dose and then administered as multiple doses for 7 days. The effect of food on the safety, tolerability and pharmacokinetics of the ABT-072 tablet will also be evaluated.

DETAILED DESCRIPTION:
The study consists of two substudies. Substudy 1 is a two-period, single ascending dose (SAD) and multiple ascending dose (MAD) blinded, randomized, placebo-controlled, non-fasting study. Designated groups that participate in Period 1 (SAD) will also participate in Period 2 (MAD). Substudy 2 is an open-label, randomized two-period, crossover study to examine the effect of food on the pharmacokinetics of ABT 072.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy subjects, non-childbearing females included.

Exclusion Criteria:

* Use of any medications (prescription and over-the-counter), vitamins, or herbal supplements within the 2-week period prior to the first dose of study drug administration or within 10 half-lives of the respective medication, whichever is longer.
* Pregnant or breast-feeding female.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab).
* Positive screen for drugs of abuse, alcohol, or cotinine.
* Clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder.
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the single and multiple dose safety and tolerability of the ABT-072 tablet formulation under non-fasting conditions. | Up to 14 days post last dose.
To determine the single and multiple dose safety pharmacokinetics of the ABT-072 tablet formulation under non-fasting conditions. | 72 hours post last dose.

SECONDARY OUTCOMES:
To assess the effect of food on the pharmacokinetics of the ABT-072 tablet formulation. | 72 hours post last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 23742, Waukegan, Illinois, United States